CLINICAL TRIAL: NCT05060432
Title: A Multicenter, Open-Label, Phase I/II Study of EOS884448 (EOS-448) in Combination With Standard of Care and/or Investigational Therapies in Participants With Advanced Solid Tumors
Brief Title: Study of EOS-448 With Standard of Care and/or Investigational Therapies in Participants With Advanced Solid Tumors
Acronym: TIG-006
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iTeos Belgium SA (Industry)
Collaborators: GlaxoSmithKline (Industry); iTeos Therapeutics (Industry)
Responsible Party: Sponsor
Organization: iTeos Therapeutics (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TIG-006
Record Dates: First submitted 2021-09-06; First posted 2021-09-29 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Advanced Cancer; Lung Cancer; Head and Neck Cancer; Melanoma
Keywords: EOS884448; GSK4428859A; TIGIT; Anti-TIGIT; EOS-448; pembrolizumab; dostarlimab; inupadenant; A2A Receptor antagonist; EOS-850; EOS100850; Anti-PD-1 monoclonal antibody; belrestotug
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Melanoma | interventions — pembrolizumab; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1A - EOS-448 + pembrolizumab (Experimental): Participants will receive EOS-448 and pembrolizumab at every cycle
  Interventions: Drug: EOS-448; Drug: pembrolizumab
- Part 1B - EOS-448 + inupadenant (Experimental): Participants will receive EOS-448 at every cycle and inupadenant on an ongoing basis
  Interventions: Drug: EOS-448; Drug: inupadenant
- Part 1C - EOS-448 + inupadenant (Experimental): Participants will receive EOS-448 at every cycle and inupadenant on an ongoing basis
  Interventions: Drug: EOS-448; Drug: inupadenant
- Part 1D - EOS-448 + dostarlimab (Experimental): Participants will receive EOS-448 and dostarlimab at every cycle
  Interventions: Drug: EOS-448; Drug: Dostarlimab
- Part 1E - inupadenant HCl + dostarlimab (Experimental): Participants will receive dostarlimab at every cycle and inupadenant on an ongoing basis
  Interventions: Drug: inupadenant; Drug: Dostarlimab
- Part 1F - EOS-448 + dostarlimab + inupadenant HC (Experimental): Participants will receive EOS-448 and dostarlimab at every cycle and inupadenant on an ongoing basis
  Interventions: Drug: EOS-448; Drug: inupadenant; Drug: Dostarlimab
- Part 1G - EOS-448 + dostarlimab + chemotherapies (Experimental): Participants with 1L mNSCLC will receive EOS-448 and dostarlimab and chemotherapies at every cycle
  Interventions: Drug: EOS-448; Drug: Dostarlimab; Drug: SOC chemotherapies
- Part 2C - EOS-448 + dostarlimab (Experimental): Participants with 1L mHNSCC CPS ≥ 20 will receive EOS-448 and dostarlimab at every cycle
  Interventions: Drug: EOS-448; Drug: Dostarlimab
- Part 2D - EOS-448 + dostarlimab (Experimental): Participants with 1L mHNSCC 1 < CPS < 20 will receive EOS-448 and dostarlimab at every cycle
  Interventions: Drug: EOS-448; Drug: Dostarlimab

INTERVENTIONS:
Drug: EOS-448 — Anti-TIGIT monoclonal antibody
  Other Names: EOS884448; GSK4428859; belrestotug
  Arms: Part 1A - EOS-448 + pembrolizumab; Part 1B - EOS-448 + inupadenant; Part 1C - EOS-448 + inupadenant; Part 1D - EOS-448 + dostarlimab; Part 1F - EOS-448 + dostarlimab + inupadenant HC; Part 1G - EOS-448 + dostarlimab + chemotherapies; Part 2C - EOS-448 + dostarlimab; Part 2D - EOS-448 + dostarlimab
Drug: pembrolizumab — Anti-PD-1 monoclonal antibody
  Arms: Part 1A - EOS-448 + pembrolizumab
Drug: inupadenant — A2A receptor antagonist
  Other Names: EOS100850
  Arms: Part 1B - EOS-448 + inupadenant; Part 1C - EOS-448 + inupadenant; Part 1E - inupadenant HCl + dostarlimab; Part 1F - EOS-448 + dostarlimab + inupadenant HC
Drug: Dostarlimab — Anti-PD-1 monoclonal antibody
  Arms: Part 1D - EOS-448 + dostarlimab; Part 1E - inupadenant HCl + dostarlimab; Part 1F - EOS-448 + dostarlimab + inupadenant HC; Part 1G - EOS-448 + dostarlimab + chemotherapies; Part 2C - EOS-448 + dostarlimab; Part 2D - EOS-448 + dostarlimab
Drug: SOC chemotherapies — SOC chemotherapies in 1L mNSCLC
  Arms: Part 1G - EOS-448 + dostarlimab + chemotherapies

SUMMARY:
This is a multicenter, open-label, phase I/II basket study, evaluating the safety, tolerability, RP2D, pharmacokinetics, pharmacodynamics and antitumor activity of EOS-448 (also known as GSK4428859A or belrestotug) combined with standard of care and/or with investigational therapies in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The combinations evaluated will be:

* EOS-448 combined with pembrolizumab, an anti-PD-1 antibody
* EOS-448 combined with inupadenant an investigational adenosine A2A receptor antagonist
* EOS-448 combined with dostarlimab an anti-PD-1 antibody
* inupadenant combined with dostarlimab
* EOS-448 combined with inupadenant and dostarlimab
* EOS-448 combined with dostarlimab and standard of care chemotherapies in participants with NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed written informed consent for the trial
* Have measurable disease, per RECIST v1.1
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 or 1.
* Have adequate organ functions
* Part 1A/1B/1C/1D/1E/1F: Have histologically or cytologically confirmed advanced or metastatic solid tumor for whom no standard treatment with survival benefit is available

Part 1G (NSCLC):

* Have a histologically confirmed or cytologically confirmed previously untreated stage IV OR stage III not amenable to curative chemoradiotherapy or surgery (AJCC 8th edition) nonsquamous NSCLC OR squamous NSCLC.
* Are eligible to receive anti-PD(L)1 therapy combined with chemotherapy in first line metastatic setting

Part 2 (H&N cancer)

* Have histologically or cytologically confirmed recurrent advanced or metastatic head and neck squamous cell carcinoma considered incurable by local therapies
* PD-L1 status positive

Exclusion Criteria:

* Have received any anti-cancer therapy within 4 weeks prior to the first dose
* Have received a live vaccine within 30 days prior to the first dose
* Have known primary CNS cancer.
* Have known CNS metastases unless previously treated and well controlled for at least 1 month
* Have concomitant second malignancies unless a complete remission was achieved at least 2 years before study entry
* Have a history of Grade ≥ 2 pneumonitis, active autoimmune disease, or persistent immune-mediated toxicity caused by immune checkpoint inhibitor therapy of Grade ≥ 2
* Have toxicity (except for alopecia) related to prior anti-cancer therapy and/or surgery unless the toxicity is either resolved, returned to baseline or Grade 1, or deemed irreversible.
* Have uncontrolled or significant cardiovascular disease
* Part 1: major surgery within 3 weeks before initiating treatment
* Part 1: Have received prior radiotherapy within 2 weeks of start of study treatment
* Part 2 (H&N cancer):
* Have received prior immunotherapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Have received prior chemotherapy administered in the recurrent advanced or metastatic setting (except for systemic therapy completed > 6 months prior to screening if given as part of multimodal treatment for locally advanced disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with DLT and Adverse Events | From first study treatment administration through Day 21-28 for DLT / Up to 120 days after the last dose
Recommended Phase 2 dose (RP2D) of EOS884448 in participants with advanced solid tumors | Up to 48 weeks
Percentage of participants with Objective Response as determined by Investigator | Until disease progression - Approximately 48 months

SECONDARY OUTCOMES:
Duration of Response (DOR) | Until disease progression or death - Approximately 48 months
Disease Control Rate (DCR) | Until disease progression or death - Approximately 48 months
Progression-free-survival (PFS) | Until disease progression or death - Approximately 48 months
Mean and median Maximum concentration (Cmax) of EOS884448 at each dose level | Up to 48 weeks
Percentage of participants with anti-drug antibodies to EOS884448 | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iteos Clinical Trials, Study Director — iTeos Belgium SA
Locations (42):
- United States (2):
  - University of California San Diego, San Diego, California
  - Hackensack University Medical Center, Bergen, New Jersey
- Belgium (5):
  - GZA Ziekenhuizen campus Sint-Augustinus, Antwerp, Antwerp
  - Cliniques universitaires St Luc-UCL, Brussels
  - Jessa Ziekenhuis, Hasselt
  - UZ Leuven, Leuven
  - CHU Helora, Mons
- France (12):
  - Hôpital Saint André, Bordeaux
  - CHU Caen, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut de Cancerologie Lorraine (ICL), Nancy
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Pitié Salpêtrière, Paris
  - CHU de POITIERS, Poitiers
  - ICANS, Strasbourg
- Italy (4):
  - IDB Center-Istituto Clinico Humanitas (IRCCS), Rozzano, Milan
  - FPO-IRCCS Candiolo Cancer Insitute, Candiolo, Turin
  - Universita degli Studi di Pavia - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AUSL Della Romagna - Ospedale S. Maria delle Croci, Ravenna
- Spain (14):
  - Hospital Althaia Xarxa Assitencial de Manresa, Manresa, Catalonia
  - Hospital Universitario de Badajoz, Badajoz
  - Vall d'Hebron, Barcelona
  - Hospital Universitario de Jaen, Jaén
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz - START Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Quirón Málaga, Málaga
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
  - Fundacion Instituto Valenciano de Oncologia (IVO), Valencia
  - Consorci Hospital Gral Univ Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (5):
  - Royal Marsden Hospital (Sutton location), Sutton, Surrey
  - Addenbrooke's Hospital, Cambridge
  - Royal Marsden Hospital (London location), London
  - Hammersmith Hospital, London
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No